CLINICAL TRIAL: NCT04078477
Title: Prevention of Pressure Ulcer by Lateral Tilt Bed in Neurocritical Care
Acronym: PULAT-NC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In accordance with the interim statistical analysis conducted after 250 patients.
Sponsor: Regional Hospital Liberec (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Vera Spatenkova, MD, Ph.D., Head of Neurointensive Care Unit, Neurocenter, Regional Hospital Liberec
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHL-NICU-2019-01
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer; Neurocritical Care; Acute Brain Disease; Unconsciousness; Preventive Strategy
MeSH Terms: conditions — Pressure Ulcer; Unconsciousness | interventions — Posture

STUDY DESIGN:
Intervention Model Description: Intervention: parallel assignment. Blind for statisticians: statisticians from a different institution will only know type A or B randomization.
Who Masked: Care Provider
Masking Description: Research Randomizer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral tilt bed (Experimental): Special lateral tilt bed.
  Interventions: Other: Body positioning
- Body positioning (No Intervention): Standard NICU preventive strategy

INTERVENTIONS:
Other: Body positioning — Comparison lateral tilt bed to standard patient´s body positioning in the bed.
  Arms: Lateral tilt bed

SUMMARY:
Patient positioning is an essential part of a preventive strategy for neurocritical care patients.

The aim of the study will be to determine whether the positioning of the bed is the same or better compared to the positioning of the patient's bed in the presence of pressure ulcer.

DETAILED DESCRIPTION:
In the monocentric, intervention, prospective, randomized study, we will investigate incidence of pressure ulcer in 300 adult consecutive patients admitted to our Neurointensive Care Unit (NICU). All patients will suffer from acute primary brain disease and will be unconscious with artificial pulmonary ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Primary brain disease
* Hospitalization in JIP neurocenter
* Age> 18 years
* Unconsciousness
* Artificial pulmonary ventilation

Exclusion Criteria:

* Intracranial hypertension
* Decubitus on the skin upon admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence of pressure ulcer | Through study completion, on average every 24 weeks.
  Pressure ulcer will be evaluated in accordance with EPUAP (European Pressure Ulcer Advisory Panel)

SECONDARY OUTCOMES:
Prolonging the stay in the NICU | Through study completion, on average every 24 weeks.
  The incidence of the pressure ulcer shall prolong the patient´s NICU stay
Cost effectiveness of patient´s NICU stay | Through study completion, on average every 24 weeks.
  Therapeutic Intervention Scoring System (TISS)

CONTACTS AND LOCATIONS:
Overall Officials: Vendula Machackova, MSc., Ph.D., Study Chair — Department for Science and Reseach
Locations (1):
- Regional Hospital Liberec, Liberec, Czechia

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analysed during the current study are available from the corresponding author on reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04078477/Prot_SAP_000.pdf